CLINICAL TRIAL: NCT05282498
Title: Pathophysiologic Mechanism for MYOcarditis in COVID19 VAccinations ("MYOVAx" Study)
Acronym: MYOVAx
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: KK Women's and Children's Hospital (Other Government); Changi General Hospital (Other); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); National University Hospital, Singapore (Other); Sengkang General Hospital (Other); Ng Teng Fong General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MYOVAx
Record Dates: First submitted 2022-03-15; First posted 2022-03-16 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Myocarditis
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected for biomarker analysis and whole genome sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The coronavirus disease 2019 (COVID-19) is an ongoing pandemic which has infected more than 160 million people and caused 3.4 million deaths worldwide till May 2021. With the recent rollout of COVID-19 vaccines globally and in Singapore, reports of rare but serious cardiovascular-related side effects started to appear. Although a link between adenovirus-based vaccines (AstraZeneca ChAdOx1 and J&J Ad26.COV2.S) and cerebral venous sinus thrombosis (CVST) and immune thrombocytopenia has been widely reported, these vaccines are current not in use in Singapore. Yet, acute myocarditis and other cardiovascular symptoms has also been observed to be associated with the two mRNA-based vaccines (Pfizer-BioNTech BNT162b2 and Moderna mRNA-1273) in-use in Singapore. In Singapore acute myocarditis is of particular concern with at least 12 cases reported by the Health Services Authority (HSA). The US FDA and EU authorities have confirmed there to be an association between the mRNA vaccines and myocarditis.The study aims to (1) To study possible mechanisms of COVID-19 vaccines in causing myocarditis in patients with confirmed vaccine-associated myocarditis (2) To risk stratify for vaccine-associated myocarditis in the at-risk population of young men (3) To identify potential preventative strategies to mitigate vaccine-associated myocarditis in high-risk individuals

DETAILED DESCRIPTION:
This is a prospective cohort study of patients with confirmed COVID19 vaccine associated myocarditis (CVAM). Patients will be required to fulfil CDC criteria for probable myocarditis with an enriched subset of confirmed cases. Study team will consent patients diagnosed with probably or confirmed myocarditis based on CDC criteria. Of the criteria, all patients must have elevated cardiac troponins. Patients will need to have a prior history of COVID19 vaccination within 21 days prior to the onset of symptoms. Clinical data, blood for serology, spike protein and mRNA measurements, biomarkers including immune mediators and cytokines will be analysed. Whole genome sequencing will also be performed. Patients will also undergo cardiac MRI. Patient will have clinical follow up at month-6 and blood samples analysis will be repeated. Cardiac MRI will be repeated at month-6 for those whose initial cardiac MRI show evidence of myocarditis to evaluate for recovery.

ELIGIBILITY:
Inclusion Criteria:

1. All patients age admitted to inpatient wards of public hospitals with cardiovascular complaints of chest pain, breathlessness, and/or palpitations, who have prior COVID19 vaccination within 21 days and who meet probable or confirmed criteria for myocarditis according to CDC (Annex A).
2. All patients age presented to outpatient clinics of public hospitals with complaints of chest pain, breathlessness, and/or palpitations accompanied with rise of cardiac Troponin biomarker, who have prior COVID19 vaccination within 30 days and who meet probable or confirmed criteria for myocarditis according to CDC (Annex A).
3. Age >/= 5. Patients under age 21 will need parental consent.
4. Willing to adhere to study protocol and other study requirements
5. Provide informed consent
6. Women who are pregnant or are breastfeeding may be included but will not be offered cardiac MRI with contrast, for safety reasons.

Exclusion Criteria:

1. Known prior abnormal heart function
2. Contraindication to cardiac MRI
3. Any condition which the investigator believes will prevent adherence to study protocol

Ages: 5 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. All patients age admitted to inpatient wards of public hospitals with cardiovascular complaints of chest pain, breathlessness, and/or palpitations, who have prior COVID19 vaccination within 21 days and who meet probable or confirmed criteria for myocarditis according to CDC (Annex A).
  2. All patients age presented to outpatient clinics of public hospitals with complaints of chest pain, breathlessness, and/or palpitations accompanied with rise of cardiac Troponin biomarker, who have prior COVID19 vaccination within 30 days and who meet probable or confirmed criteria for myocarditis according to CDC (Annex A).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac MRI | Cardiac MRI should be done within 2 weeks from presentation
  Myocarditis will be grouped according to:
  i. Group 1. Patients with cardiac symptoms, elevated troponins and normal cardiac function on echo ii. Group 2. Patients with cardiac symptoms, elevated troponins </=30 times upper limit of normal range (for the individual hospital), regardless of cardiac function on echo iii. Group 3. Patients with cardiac symptoms, elevated troponins > 30 times upper limit of normal range (for the individual hospital), regardless of cardiac function on echo iv. Group 4. Myocarditis diagnosed according to CDC criteria not meeting above categories

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore